CLINICAL TRIAL: NCT07344649
Title: Turkish Validation of the Nijmegen Questionnaire in COPD
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: Nijmegen&TR
Record Dates: First submitted 2026-01-01; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Administration of validated self-reported questionnaires (Nijmegen Questionnaire, CAT, mMRC, HADS, Dyspnea-12)

SUMMARY:
Dysfunctional breathing is a common and clinically relevant problem in patients with chronic obstructive pulmonary disease (COPD), contributing to increased dyspnea perception, reduced exercise tolerance, and impaired quality of life. The Nijmegen Questionnaire (NQ) is a widely used symptom-based instrument for screening dysfunctional breathing; however, a validated Turkish version for patients with COPD is currently unavailable.

This observational methodological study aims to translate, culturally adapt, and evaluate the validity and reliability of the Turkish version of the Nijmegen Questionnaire (NQ-TR) in individuals with stable COPD.

DETAILED DESCRIPTION:
This single-center observational study will be conducted in patients with clinically stable COPD. The study consists of two main phases: (1) translation and cultural adaptation of the Nijmegen Questionnaire following international guidelines for patient-reported outcome measures, and (2) psychometric evaluation of the Turkish version in a COPD population.

The translation process includes forward translation, reconciliation, back-translation, developer review, cognitive debriefing with patients, and final proofreading. After completion of the linguistic adaptation, the NQ-TR will be administered to eligible participants at baseline and repeated after one week in clinically stable individuals to assess test-retest reliability.

Construct validity will be evaluated using exploratory and confirmatory factor analyses. Convergent validity will be assessed by examining correlations between NQ-TR scores and established clinical measures, including the COPD Assessment Test (CAT), Modified Medical Research Council (mMRC) Dyspnea Scale, Hospital Anxiety and Depression Scale (HADS), and Dyspnea-12 (D-12). Internal consistency, test-retest reliability, and measurement stability will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosis of COPD confirmed according to GOLD criteria
* Clinically stable disease (no acute exacerbation or hospitalization within the last 4 weeks)
* Ability to read and understand Turkish
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Acute COPD exacerbation or respiratory infection within the previous 4 weeks
* Presence of severe cardiac, neurological, or systemic disease affecting questionnaire responses
* Coexisting pulmonary conditions such as bronchiectasis, lung cancer, prior pulmonary tuberculosis, pleural disease, or history of lung surgery
* Moderate to severe cognitive impairment or communication difficulties
* Severe visual or hearing impairment preventing questionnaire completion
* Pregnancy
* Refusal to participate or withdrawal during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 years and older with a confirmed diagnosis of chronic obstructive pulmonary disease (COPD) according to GOLD criteria. Eligible participants are clinically stable patients attending the pulmonology outpatient clinic of a tertiary care hospital, with no acute exacerbation or hospitalization within the previous four weeks. All participants are Turkish-speaking, able to complete self-reported questionnaires, and provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Turkish version of the Nijmegen Questionnaire (NQ-TR) | Baseline and 1 week
  The Nijmegen Questionnaire is a validated self-report instrument used to assess symptoms related to dysfunctional breathing and hyperventilation. It consists of 16 items evaluating the frequency of respiratory and non-respiratory symptoms, with higher total scores indicating greater symptom severity. In this study, the Turkish-validated version of the Nijmegen Questionnaire (NQ-TR) will be used to evaluate dysfunctional breathing symptoms in participants.

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) | Baseline
  The COPD Assessment Test (CAT) is a validated, patient-completed questionnaire designed to assess the impact of chronic obstructive pulmonary disease (COPD) on health status. It consists of 8 items covering symptoms, activity limitation, and overall well-being, with total scores ranging from 0 to 40. Higher scores indicate a greater impact of COPD on health status. In this study, the Turkish-validated version of the COPD Assessment Test (CAT) will be used to evaluate disease-related symptom burden and health status in participants with COPD.
Modified Medical Research Council (mMRC) Dyspnea Scale | Baseline
  The Modified Medical Research Council (mMRC) Dyspnea Scale is a widely used, validated scale for assessing the severity of perceived breathlessness related to physical activity in individuals with chronic respiratory diseases. The scale grades dyspnea from 0 to 4, with higher grades indicating greater functional limitation due to breathlessness. In this study, the Turkish-validated version of the Modified Medical Research Council (mMRC) Dyspnea Scale will be used to assess dyspnea severity in participants.
Dyspnea-12 (D-12) Scale | Baseline
  The Dyspnea-12 (D-12) Scale is a validated patient-reported outcome measure designed to assess both the physical and affective components of breathlessness. It consists of 12 items, with total scores ranging from 0 to 36, where higher scores indicate greater dyspnea severity. In this study, the Turkish-validated version of the Dyspnea-12 (D-12) Scale will be used to evaluate the multidimensional severity of dyspnea in participants.
Hospital Anxiety and Depression Scale (HADS) | Baseline
  The Hospital Anxiety and Depression Scale (HADS) is a validated self-report questionnaire designed to assess symptoms of anxiety and depression in individuals with physical health conditions. It consists of 14 items divided into two subscales: anxiety (HADS-A) and depression (HADS-D), each comprising 7 items, with subscale scores ranging from 0 to 21. Higher scores indicate greater psychological distress. In this study, the Turkish-validated version of the Hospital Anxiety and Depression Scale (HADS) will be used to evaluate anxiety and depression levels in participants.